CLINICAL TRIAL: NCT03420391
Title: Effects of Photobiomodulation Therapy (PBMT) on Muscular Performance and Recovery in Different Time-points
Brief Title: PBMT on Muscular Performance and Recovery in Different Time-points
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); University of Bergen (Other)
Responsible Party: Principal Investigator, Ernesto Cesar Pinto Leal Junior, Full professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 113553
Record Dates: First submitted 2018-01-20; First posted 2018-02-05 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Phototherapy
Keywords: phototherapy; performance; muscular recovery; photobiomodulation therapy; time-window
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Sixty participants will be enrolled in the study. Participants will be randomized in six groups:
  Control: Participants will receive no intervention; Placebo: Participants will receive placebo PBMT; 5 minutes: Participants will perform the eccentric exercise protocol 5 minutes after PBMT.
  3 hours: Participants will perform the eccentric exercise protocol 3 hours after PBMT.
  6 hours: Participants will perform the eccentric exercise protocol 6 hours after PBMT.
  24 hours: Participants will perform the eccentric exercise protocol 24 hours after PBMT.
  Assessments will be performed at baseline, after 1 minute, 1 hour, 24 and 48 hours after the end of exercise protocol.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Placebo PBMT (Placebo Comparator): Participants will be treated with placebo PBMT in different time-points before the eccentric exercise protocol (5 minutes, 3 hours, 6 hours or 24 hours). Assessments will be performed at baseline, 1 minute, 1 hour, 24 and 48 hours after the end of exercise protocol.
  Interventions: Device: Photobiomodulation Therapy (PBMT)
- 5 Minutes (Active Comparator): Participants will be performed the eccentric exercise protocol 5 minutes after PBMT.
  Assessments will be performed at baseline, 1 minute, 1 hour, 24 and 48 hours after the end of exercise protocol.
  Interventions: Device: Photobiomodulation Therapy (PBMT)
- 3 Hours (Active Comparator): 3 hours: Participants will be performed the eccentric exercise protocol 3 hours after PBMT.
  Assessments will be performed before at baseline, 1 minute, 1 hour and 24, 48 hours after the end of exercise protocol.
  Interventions: Device: Photobiomodulation Therapy (PBMT)
- 6 Hours (Active Comparator): 6 hours: Participants will be performed the eccentric exercise protocol 6 hours after PBMT.
  Assessments will be performed at baseline, 1 minute, 1 hour, 24 and 48 hours after the end of exercise protocol.
  Interventions: Device: Photobiomodulation Therapy (PBMT)
- 24 hours (Active Comparator): 24 hours: Participants will be performed the eccentric exercise protocol 24 hours after PBMT. Assessments will be performed before at baseline, 1 minute, 1 hour, 24 and 48 hours after the end of exercise protocol.
  Interventions: Device: Photobiomodulation Therapy (PBMT)
- Control (No Intervention): Participants will not receive intervention. Assessments will be performed at baseline, 1 minute, 1 hour, 24 and 48 hours after the end of exercise protocol.

INTERVENTIONS:
Device: Photobiomodulation Therapy (PBMT) — Phototherapy device - Multi Radiance Medical® (Solon, OH, EUA)
  Arms: 24 hours; 3 Hours; 5 Minutes; 6 Hours; Placebo PBMT

SUMMARY:
Recent studies with photobiomodulation therapy (PBMT) have shown positive results delaying skeletal muscle fatigue and improving the status of biochemical markers related to skeletal muscle damage when these therapies were applied before exercise. The aim of this project is to verify the effects of PBMT in improvement of skeletal muscle performance and skeletal muscle recovery in healthy male subjects. This project aim also to validate the concept that simultaneous use of three wavelengths and light sources lead to optimized action independently of time-window between irradiation and the exercise.

DETAILED DESCRIPTION:
This is a randomized, triple-blinded, placebo-controlled trial. Sixty healthy untrained male subjects will be randomly allocated to six experimental groups: Placebo, Control, PBMT 5 mins, PBMT 3h, PBMT 6h and PBMT 24 hours. PBMT will be applied precisely two minutes after baseline MVC test. Then, after five minutes, 3, 6 hours or 1 day (24 hours) of PBMT the eccentric exercise protocol will be performed. We will analyze maximum voluntary contraction (MVC), creatine kinase (CK) activity and delayed onset muscle soreness (DOMS). Assessments will be performed at baseline, immediately after (1 minute), 1 hour, 24 and 48 hours after the eccentric exercise protocol.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* not athletes or who engage in physical activity at most once a week
* Individuals should not present a history of musculoskeletal injury in the hip and knee regions in the two months prior to the studies
* they should not be using pharmacological agents and / or nutritional supplements
* They must attend 100% of the data collections.

Exclusion Criteria:

* Individuals who do not meet the criteria mentioned above or who present musculoskeletal damage during collection were excluded from the study.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2019-07-19 (Actual); Study Completion 2019-07-19 (Actual)

PRIMARY OUTCOMES:
Torque peak / maximum voluntary contraction - MVC | 1 minute, 1 hour, 24 and 48 hours after the end of exercise protocol.
  Assessment was performed in the isokinetic dynamometer (System 4, Biodex®, USA)

SECONDARY OUTCOMES:
Delayed onset muscle soreness (DOMS) | 1 minute, 1 hour, 24 and 48 hours after the end of exercise protocol.
  Assessment was performed through visual analogue scale (VAS). A visual analogue scale (VAS) of 100 mm was used as a self-rating of volunteers DOMS intensity, with assistance of a blinded researcher, where "0" corresponds to no pain and 100mm corresponds to the worst pain possible.
Biochemical marker of muscle damage | 1 minute, 1 hour, 24 and 48 hours after the end of exercise protocol.
  Analysis of Creatine Kinase (CK) levels

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Nove de Julho, São Paulo, Brazil

REFERENCES:
- [Derived] Leal-Junior ECP, de Oliveira MFD, Joensen J, Stausholm MB, Bjordal JM, Tomazoni SS. What is the optimal time-response window for the use of photobiomodulation therapy combined with static magnetic field (PBMT-sMF) for the improvement of exercise performance and recovery, and for how long the effects last? A randomized, triple-blinded, placebo-controlled trial. BMC Sports Sci Med Rehabil. 2020 Oct 19;12:64. doi: 10.1186/s13102-020-00214-8. eCollection 2020. PMID 33088573